CLINICAL TRIAL: NCT04664153
Title: A PHASE 2A, RANDOMIZED, DOUBLE BLIND, VEHICLE CONTROLLED, PARALLEL GROUP STUDY TO ASSESS THE EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-07038124 OINTMENT FOR 6 WEEKS IN PARTICIPANTS WITH MILD TO MODERATE ATOPIC DERMATITIS OR PLAQUE PSORIASIS
Brief Title: Study To Assess Efficacy, Safety, Tolerability And Pharmacokinetics Of PF-07038124 Ointment In Participants With Atopic Dermatitis Or Plaque Psoriasis
Acronym: EMPORIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3941002; 2020-003977-23 (EudraCT Number)
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis; Plaque Psoriasis
Keywords: atopic dermatitis, plaque psoriasis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- atopic dermatitis - PF-07038124 ointment (Experimental)
  Interventions: Drug: PF-07038124 ointment
- atopic dermatitis - vehicle ointment (Placebo Comparator)
  Interventions: Drug: Vehicle ointment
- plaque psoriasis - PF-07038124 ointment (Experimental)
  Interventions: Drug: PF-07038124 ointment
- plaque psoriasis - vehicle ointment (Experimental)
  Interventions: Drug: Vehicle ointment

INTERVENTIONS:
Drug: PF-07038124 ointment — PF-07038124 ointment at 0.01% with QD dosing for 6 weeks
  Arms: atopic dermatitis - PF-07038124 ointment; plaque psoriasis - PF-07038124 ointment
Drug: Vehicle ointment — Vehicle ointment with QD dosing for 6 weeks
  Arms: atopic dermatitis - vehicle ointment; plaque psoriasis - vehicle ointment

SUMMARY:
This study is being conducted to provide data on efficacy, safety, tolerability and PK of PF-07038124 ointment versus vehicle control in the treatment of mild to moderate AD and mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Atopic Dermatitis (AD): Have been diagnosed with AD for at least 3 months; Have an Investigator's Global Assessment (IGA) score of 2 (mild), or 3 (moderate); Have AD covering 5% to 20% (inclusive) of BSA.
* Plaque psoriasis: Have been diagnosed with plaque psoriasis (psoriasis vulgaris) for at least 6 months; Have a Physician Global Assessment (PGA) score of 2 (mild), or 3 (moderate); Having plaque psoriasis covering 5% to 15% (inclusive) of BSA.

Exclusion Criteria:

* Presence of skin comorbidities that would interfere with study assessment or response to treatment.
* Current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurological disease.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (15):
  - First OC Dermatology, Fountain Valley, California
  - Renaissance Research and Medical Group, Cape Coral, Florida
  - Olympian Clinical Research, Clearwater, Florida
  - Moonshine Research Center, Inc., Doral, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Center for Clinical Studies, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Henry Ford Medical Center, New Center One, Detroit, Michigan
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Memphis, Tennessee
  - studies in Dermatology, LLC, Cypress, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas
- Australia (2):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Emeritus Research, Camberwell, Victoria
- Canada (5):
  - Dermatrials Research Inc., Hamilton, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec
- Poland (7):
  - NZOZ Specjalistyczny Osrodek Dermatologiczny DERMAL, Bialystok
  - Mazowieckie Centrum Badań Klinicznych, Grodzisk Mazowiecki
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Kliniczny Szpital Wojewódzki nr 1 im. F. Chopina w Rzeszowie, Rzeszów
  - ETG Warszawa, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Eichenfield LF, Tarabar S, Forman S, Garcia-Bello A, Feng G, Fetterly G, Mahling P, Peeva E, Vincent MS, Chandra DE. Efficacy and Safety of PF-07038124 in Patients With Atopic Dermatitis and Plaque Psoriasis: A Randomized Clinical Trial. JAMA Dermatol. 2024 Feb 1;160(2):156-163. doi: 10.1001/jamadermatol.2023.4990. PMID 38117526
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3941002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 152 participants were screened for this study and 104 participants were assigned to study treatment (70 for atopic dermatitis [AD] group and 34 for plaque psoriasis group).
Groups:
- AD Vehicle Once Daily (QD): Participants in AD group received vehicle ointment in 60 g tube with QD dosing beginning on Day 1 through the final dose at Week 6 visit.
- AD PF-07038124 0.01% QD: Participants in AD group received PF-07038124 ointment at 0.01% in 60 g tube with QD dosing beginning on Day 1 through the final dose at Week 6 visit.
- Psoriasis Vehicle QD: Participants in plaque psoriasis group received vehicle ointment in 60 g tube with QD dosing beginning on Day 1 through the final dose at Week 6 visit.
- Psoriasis PF-07038124 0.01% QD: Participants in plaque psoriasis group received PF-07038124 ointment at 0.01% in 60 g tube with QD dosing beginning on Day 1 through the final dose at Week 6 visit.
Period: Overall Study
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Started | 34 | 36 | 17 | 17
Completed | 27 | 33 | 13 | 15
Not Completed | 7 | 3 | 4 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 2
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD | Total
Number analyzed (Participants) | 34 | 36 | 17 | 17 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 36.1 (13.93) | 41.4 (16.61) | 51.2 (10.83) | 51.8 (12.32) | 43.0 (15.44)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 25 | 23 | 4 | 4 | 56
  45-64 years | 9 | 8 | 12 | 10 | 39
  >=65 years | 0 | 5 | 1 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 7 | 7 | 55
  Male | 13 | 16 | 10 | 10 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 7 | 5 | 31
  Not Hispanic or Latino | 26 | 25 | 10 | 12 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 29 | 17 | 16 | 87
  Black or African American | 8 | 5 | 0 | 0 | 13
  Asian | 1 | 2 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 6 for AD Participants
Description: EASI evaluated severity of participants' AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Week 6
Population: Analysis population included all participants who received at least 1 dose of study treatment. For this outcome measure (OM), data collection was not planned for the 2 arms of Psoriasis Vehicle QD and Psoriasis PF-07038124 0.01% QD.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36
Percent Change | -35.5 [-48.95 to -22.03] | -74.9 [-88.81 to -61.06]
Statistical Analysis 1: Comparison: AD Vehicle Once Daily (QD) vs AD PF-07038124 0.01% QD; Test type: Superiority; p = 0.0004, t-test, 1 sided; Mean Difference (Final Values) = -39.4, 90% CI 2-sided [-58.76 to -20.12], Standard Error of Mean 11.74

2. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 6 for Plaque Psoriasis Participants
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0= 0% to 6= 90-100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease, where higher scores = greater severity of psoriasis.
Time Frame: Baseline, Week 6
Population: Analysis population included all participants who received at least 1 dose of study treatment. For this OM, data collection was not planned for the 2 arms of AD Vehicle QD and AD PF-07038124 0.01% QD.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a Scale
Arm/Group | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 17 | 17
Units on a Scale | 0.1 [-1.47 to 1.68] | -4.8 [-6.21 to -3.37]
Statistical Analysis 1: Comparison: Psoriasis Vehicle QD vs Psoriasis PF-07038124 0.01% QD; Test type: Superiority; p < 0.0001, t-test, 1 sided; Mean Difference (Final Values) = -4.9, 90% CI 2-sided [-7.02 to -2.77], Standard Error of Mean 1.29

3. Secondary Outcome: Percentage of AD Participants Achieving Investigator's Global Assessment (IGA) Score of Clear (0) or Almost Clear (1) (on a 5-Point Scale) and a Reduction From Baseline of >=2 Points at Week 6
Description: IGA assessed severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared-light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. In this OM, percentages of participants with an IGA score of 0 or 1 and a reduction of >=2 from Baseline in IGA score are reported.
Time Frame: Baseline, Week 6
Population: Analysis population included all participants who received at least 1 dose of study treatment. For this OM, data collection was not planned for the 2 arms of Psoriasis Vehicle QD and Psoriasis PF-07038124 0.01% QD.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36
Percentage of Participants | 8.8 [3.3 to 19.7] | 44.4 [30.2 to 59.1]

4. Secondary Outcome: Percentage of AD Participants Achieving EASI 75 (75% Improvement From Baseline) at Weeks 1, 2, 4, 6 and Follow-up (FUP)/End of Study (EOS)
Description: EASI evaluated severity of participants' AD based on severity of AD clinical signs and % of BSA affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD. EASI 75 response was defined as at least a 75 percent (%) reduction in EASI relative to Baseline.
Time Frame: Baseline, Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36
Percentage of Participants
  Week 1 | 0 [0.0 to 8.0] | 8.3 [3.1 to 18.9]
  Week 2: number analyzed (Participants) | 33 | 36
  Week 2 | 0 [0.0 to 8.2] | 27.8 [15.9 to 40.9]
  Week 4 | 11.8 [5.2 to 24.3] | 33.3 [21.3 to 47.0]
  Week 6 | 20.6 [11.3 to 34.9] | 61.1 [47.0 to 74.6]
  FUP/EOS | 8.8 [3.3 to 19.7] | 44.4 [30.2 to 59.1]

5. Secondary Outcome: Percentage of AD Participants Having >=4 Points of Reduction in Weekly Averages of Peak Pruritus Numerical Rating Scale (PP-NRS) From Baseline at Weeks 1, 2, 4 and 6
Description: The PP-NRS was a daily patient-reported assessment of intensity of pruritus on an 11-point numerical rating scale, ranging from 0 ('No Itch) to 10 ('Worst Itch Imaginable') with a 24 hour recall period. For the PP-NRS score, baseline was defined as the average of all values recorded between Day -7 and Day -1. In this OM, percentages of AD participants with >=4 points of reduction in weekly averages of PP-NRS from baseline are reported (percentage based on number of participants with baseline >=4).
Time Frame: Baseline, Weeks 1, 2, 4 and 6
Population: Analysis population included all participants who received at least 1 dose of study treatment with PP-NRS baseline >=4. For this OM, data collection was not planned for the 2 arms of Psoriasis Vehicle QD and Psoriasis PF-07038124 0.01% QD.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36
Percentage of Participants
  Week 1: number analyzed (Participants) | 29 | 34
  Week 1 | 0 [0.0 to 9.4] | 8.8 [3.3 to 19.7]
  Week 2: number analyzed (Participants) | 29 | 34
  Week 2 | 3.4 [0.4 to 14.5] | 23.5 [12.3 to 37.7]
  Week 4: number analyzed (Participants) | 29 | 34
  Week 4 | 6.9 [1.8 to 20.0] | 41.2 [26.9 to 56.7]
  Week 6: number analyzed (Participants) | 29 | 34
  Week 6 | 13.8 [6.2 to 27.9] | 41.2 [26.9 to 56.7]

6. Secondary Outcome: Change From Baseline in EASI Total Score at Weeks 1, 2, 4, 6 and FUP/EOS for AD Participants
Description: EASI evaluated severity of participants' AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of BSA affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 3
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a Scale
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36
Units on a Scale
  Week 1 | -1.7 [-2.59 to -0.85] | -3.4 [-4.28 to -2.59]
  Week 2: number analyzed (Participants) | 30 | 36
  Week 2 | -2.4 [-3.42 to -1.45] | -5.6 [-6.51 to -4.66]
  Week 4: number analyzed (Participants) | 28 | 35
  Week 4 | -2.5 [-3.63 to -1.31] | -7.0 [-8.06 to -5.90]
  Week 6: number analyzed (Participants) | 30 | 34
  Week 6 | -3.3 [-4.59 to -1.93] | -8.2 [-9.39 to -6.94]
  FUP/EOS: number analyzed (Participants) | 27 | 32
  FUP/EOS | -2.8 [-4.26 to -1.39] | -6.9 [-8.19 to -5.54]

7. Secondary Outcome: Percentage of AD Participants Achieving IGA Score of Clear (0) or Almost Clear (1) at Weeks 1, 2, 4, 6 and FUP/EOS
Description: IGA assessed severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. In this OM, percentages of participants with an IGA score of 0 or 1 are reported.
Time Frame: Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36
Percentage of Participants
  Week 1 | 2.9 [0.3 to 12.3] | 11.1 [4.9 to 22.9]
  Week 2: number analyzed (Participants) | 33 | 36
  Week 2 | 9.1 [3.4 to 20.2] | 36.1 [22.9 to 50.0]
  Week 4 | 14.7 [7.3 to 26.9] | 44.4 [30.2 to 59.1]
  Week 6 | 17.6 [8.0 to 30.7] | 52.8 [38.0 to 67.2]
  FUP/EOS | 5.9 [1.6 to 16.9] | 38.9 [25.4 to 53.0]

8. Secondary Outcome: Percentage of Psoriasis Participants With Physician Global Assessment (PGA) Score Clear (0) or Almost Clear (1) (on a 5-Point Scale) and >=2 Points Improvement From Baseline at Week 6
Description: The PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). In this OM, percentages of participants with a PGA score of 0 or 1 and an improvement of >=2 from Baseline in PGA score are reported.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 17 | 17
Percentage of Participants | 5.9 [0.6 to 22.5] | 17.6 [6.7 to 36.4]

9. Secondary Outcome: Percentage of Psoriasis Participants Achieving PASI 75 (75% or Greater Improvement From Baseline) at Weeks 1, 2, 4, 6 and FUP/EOS
Description: The PASI quantified the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. PASI was a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score could vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least a 75 percent (%) reduction in PASI relative to Baseline.
Time Frame: Baseline, Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 17 | 17
Percentage of Participants
  Week 1 | 0 [0.0 to 14.0] | 5.9 [0.6 to 22.5]
  Week 2 | 0 [0.0 to 14.0] | 5.9 [0.6 to 22.5]
  Week 4 | 0 [0.0 to 14.0] | 17.6 [6.7 to 36.4]
  Week 6 | 5.9 [0.6 to 22.5] | 35.3 [17.5 to 56.8]
  FUP/EOS | 0 [0.0 to 14.0] | 23.5 [10.7 to 43.2]

10. Secondary Outcome: Percentage of Psoriasis Participants Who Achieved a Psoriasis Symptoms Inventory (PSI) Score of 0 (Not at All) or 1 (Mild) on Every Item at Weeks 1, 2, 4, 6 and FUP/EOS
Description: PSI was a self-administered 8 item questionnaire that measured the severity of psoriasis symptoms over the past 24 hours and the past 7 days. The measure included concepts of itch, pain, burning, stinging, cracking, scaling, flaking, and redness. Participants were asked to respond to each item using a 5 point Likert response scale: 0: not all severe, 1: mild, 2: moderate, 3: severe and 4: very severe. In this OM, percentages of participants with a PSI score of 0 or 1 on every item at weeks 1, 2, 4, 6 and FUP/EOS are reported.
Time Frame: Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 17 | 17
Percentage of Participants
  Week 1 | 0 [0.0 to 14.0] | 11.8 [3.2 to 31.1]
  Week 2: number analyzed (Participants) | 17 | 16
  Week 2 | 5.9 [0.6 to 22.5] | 18.8 [7.1 to 39.1]
  Week 4: number analyzed (Participants) | 17 | 16
  Week 4 | 23.5 [10.7 to 43.2] | 43.8 [23.5 to 66.7]
  Week 6 | 29.4 [14.0 to 50.0] | 58.8 [36.4 to 77.5]
  FUP/EOS | 41.2 [22.5 to 63.6] | 41.2 [22.5 to 63.6]

11. Secondary Outcome: Change From Baseline in PASI Scores at Weeks 1, 2, 4 and FUP/EOS
Description: as for outcome 2
Time Frame: Baseline, Weeks 1, 2, 4 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a Scale
Arm/Group | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 17 | 17
Units on a Scale
  Week 1 | -0.6 [-1.23 to 0.03] | -1.9 [-2.50 to -1.24]
  Week 2 | -0.7 [-1.51 to 0.11] | -3.2 [-3.97 to -2.35]
  Week 4: number analyzed (Participants) | 16 | 17
  Week 4 | -0.1 [-1.49 to 1.19] | -4.1 [-5.44 to -2.80]
  FUP/EOS: number analyzed (Participants) | 13 | 15
  FUP/EOS | 0.2 [-1.59 to 1.97] | -3.7 [-5.35 to -2.00]

12. Secondary Outcome: Percent Change From Baseline in PASI Scores at Weeks 1, 2, 4, 6 and FUP/EOS
Description: as for outcome 2
Time Frame: Baseline, Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 17 | 17
Percent Change
  Week 1 | -6.8 [-15.28 to 1.78] | -25.6 [-34.11 to -17.04]
  Week 2 | -9.0 [-19.14 to 1.09] | -37.8 [-47.92 to -27.68]
  Week 4: number analyzed (Participants) | 16 | 17
  Week 4 | -9.0 [-22.73 to 4.73] | -49.4 [-62.93 to -35.79]
  Week 6: number analyzed (Participants) | 14 | 17
  Week 6 | -5.4 [-21.35 to 10.65] | -58.1 [-73.52 to -42.70]
  FUP/EOS: number analyzed (Participants) | 13 | 15
  FUP/EOS | -8.4 [-27.02 to 10.25] | -45.6 [-63.02 to -28.10]

13. Secondary Outcome: Percentage of Psoriasis Participants With PGA Score Clear (0) or Almost Clear (1) at Weeks 1, 2, 4, 6 and FUP/EOS
Description: The PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). In this OM, percentages of participants with a PGA score of 0 or 1 are reported.
Time Frame: Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 17 | 17
Percentage of Participants
  Week 1 | 0 [0.0 to 14.0] | 11.8 [3.2 to 31.1]
  Week 2 | 0 [0.0 to 14.0] | 17.6 [6.7 to 36.4]
  Week 4 | 0 [0.0 to 14.0] | 23.5 [10.7 to 43.2]
  Week 6 | 5.9 [0.6 to 22.5] | 23.5 [10.7 to 43.2]
  FUP/EOS | 11.8 [3.2 to 31.1] | 17.6 [6.7 to 36.4]

14. Secondary Outcome: Percent Change From Baseline in Affected Body Surface Area (BSA) at Weeks 1, 2, 4, 6 and FUP/EOS
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranges from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Baseline, Weeks 1, 2, 4, 6 and FUP/EOS (28-35 days post-last dose)
Population: Analysis population included all participants who received at least 1 dose of study treatment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36 | 17 | 17
Percent Change
  Week 1 | -6.6 [-13.56 to 0.44] | -20.2 [-27.01 to -13.44] | 2.5 [-5.50 to 10.49] | -14.5 [-22.46 to -6.56]
  Week 2: number analyzed (Participants) | 30 | 36 | 17 | 17
  Week 2 | -10.5 [-19.71 to -1.27] | -32.2 [-40.83 to -23.62] | 7.2 [-2.68 to 17.17] | -13.8 [-23.70 to -3.91]
  Week 4: number analyzed (Participants) | 28 | 35 | 16 | 17
  Week 4 | -2.9 [-15.80 to 9.94] | -43.9 [-55.73 to -32.00] | 19.8 [3.80 to 35.79] | -24.7 [-40.52 to -8.89]
  Week 6: number analyzed (Participants) | 30 | 34 | 14 | 17
  Week 6 | -4.9 [-23.07 to 13.28] | -61.2 [-78.01 to -44.42] | 29.0 [4.46 to 53.46] | -32.6 [-56.32 to -8.84]
  FUP/EOS: number analyzed (Participants) | 27 | 32 | 13 | 15
  FUP/EOS | -5.1 [-20.70 to 10.56] | -48.7 [-63.05 to -34.27] | 15.8 [-12.26 to 43.76] | -31.9 [-58.60 to -5.21]

15. Secondary Outcome: Number of Participants With All-Causality Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation where participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state. An SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or resulted in congenital anomaly/birth defect.
Time Frame: Day 1 through Week 6
Population: Analysis population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36 | 17 | 17
Participants
  Participants With All-Causality TEAEs | 9 | 9 | 6 | 3
  Participants With All-Causality SAEs | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-defined Criteria
Description: Abnormality in vital signs: increase and decrease of change of supine diastolic blood pressure from baseline >=20 mmHg, supine systolic blood pressure <90 mmHg, and increase in change of supine systolic blood pressure from baseline >=30 mmHg.
Time Frame: Day 1 through Week 6
Population: Analysis population included all participants evaluated against criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36 | 17 | 16
Participants
  Change of Supine Diastolic Blood Pressure >=20 mmHg Increase | 2 | 1 | 0 | 2
  Change of Supine Diastolic Blood Pressure >=20 mmHg Decrease | 1 | 0 | 0 | 0
  Value of Supine Systolic Blood Pressure <90 mmHg | 0 | 0 | 0 | 1
  Change of Supine Systolic Blood Pressure >=30 mmHg Increase | 1 | 1 | 1 | 0

17. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-defined Criteria
Description: ECG abnormalities criteria included: value of PR interval >=300 msec, percent change of PR interval >=25/50% and change of corrected QT interval using Fridericia's Formula (QTcF) >=30 msec and <60 msec.
Time Frame: Day 1 through Week 6
Population: Analysis population included all participants evaluated against criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 27 | 33 | 13 | 15
Participants
  Value of PR Interval >=300 msec | 0 | 1 | 0 | 0
  Percent Change of PR Interval >=25/50% | 0 | 0 | 1 | 0
  Change of Corrected QT Interval Using Fridericia's Formula (QTcF) >=30 msec and <60 msec | 3 | 0 | 0 | 1

18. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]).
Time Frame: Day 1 through Week 6
Population: Analysis population included participants with at least 1 observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36 | 17 | 17
Participants
  Hemoglobin <0.8 × LLN | 0 | 1 | 0 | 0
  Ery. Mean Corpuscular Volume <0.9 × LLN | 0 | 1 | 0 | 0
  Ery. Mean Corpuscular Hemoglobin <0.9 × LLN | 0 | 1 | 0 | 0
  Leukocytes >1.5 × ULN | 0 | 0 | 0 | 1
  Lymphocytes <0.8 × LLN | 1 | 0 | 0 | 0
  Lymphocytes >1.2 × ULN | 0 | 1 | 0 | 0
  Lymphocytes/Leukocytes <0.8 × LLN | 3 | 2 | 2 | 1
  Lymphocytes/Leukocytes >1.2 × ULN | 1 | 0 | 0 | 0
  Neutrophils <0.8 × LLN | 2 | 0 | 0 | 0
  Neutrophils >1.2 × ULN | 0 | 1 | 1 | 1
  Neutrophils/Leukocytes <0.8 × LLN | 1 | 1 | 0 | 0
  Basophils/Leukocytes >1.2 × ULN | 0 | 0 | 0 | 1
  Eosinophils >1.2 × ULN | 2 | 1 | 0 | 1
  Eosinophils/Leukocytes >1.2 × ULN | 3 | 4 | 0 | 1
  Monocytes >1.2 × ULN | 0 | 1 | 0 | 0
  Monocytes/Leukocytes >1.2 × ULN | 0 | 2 | 0 | 1
  Potassium >1.1 × ULN | 0 | 0 | 2 | 1
  Bicarbonate <0.9 × LLN | 2 | 0 | 1 | 0
  Glucose >1.5 × ULN | 2 | 3 | 4 | 1
  Fibrinogen >1.25 × ULN | 3 | 11 | 4 | 1
  URINE Glucose >=1 | 2 | 2 | 1 | 0
  Ketones >=1 | 0 | 2 | 1 | 3
  URINE Protein >=1 | 1 | 0 | 0 | 1
  URINE Hemoglobin >=1 | 4 | 4 | 2 | 2
  URINE Bilirubin >=1 | 0 | 0 | 1 | 0
  Nitrite >=1 | 2 | 0 | 0 | 0
  Leukocyte Esterase >=1 | 3 | 9 | 5 | 3
  URINE Erythrocytes (/HPF) >=20: number analyzed (Participants) | 15 | 16 | 12 | 8
  URINE Erythrocytes (/HPF) >=20 | 2 | 1 | 0 | 3
  URINE Leukocytes (/HPF) >=20: number analyzed (Participants) | 18 | 20 | 13 | 10
  URINE Leukocytes (/HPF) >=20 | 0 | 1 | 2 | 2
  Hyaline Casts (/LPF) >1: number analyzed (Participants) | 0 | 4 | 2 | 0
  Hyaline Casts (/LPF) >1 | 0 | 3 | 2 | 0

19. Secondary Outcome: Number of Participants With Different Severity Grades in Skin Tolerability at Day 1, Weeks 1, 2, 4, 6, Early Termination (ET) and FUP
Description: The investigator or designee assessed tolerability at the site of investigational product application (pre-dose and immediately post-dose). This assessment focused on the treated non-lesional skin using the scale: none = no evidence of local intolerance; mild = minimal erythema and/or oedema, slight glazed appearance; moderate = definite erythema and/or oedema with peeling and/or cracking but needs no adaptation of posology; severe (to be reported as an AE) = erythema, oedema glazing with fissures, few vesicles or papules: consider removing topical agent (if still in place); very severe (to be reported as an AE) = strong reaction spreading beyond the treated area, bullous reaction, erosions: removal of topical agent (if still in place).
Time Frame: Day 1, Weeks 1, 2, 4, 6, ET and FUP (28-35 days post-last dose)
Population: Analysis population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
Number analyzed (Participants) | 34 | 36 | 17 | 17
Participants
  Day 1 None | 33 | 35 | 17 | 17
  Day 1 Mild | 0 | 1 | 0 | 0
  Day 1 Moderate | 1 | 0 | 0 | 0
  Day 1 Severe | 0 | 0 | 0 | 0
  Day 1 Very Severe | 0 | 0 | 0 | 0
  Week 1 None | 25 | 33 | 17 | 16
  Week 1 Mild | 4 | 3 | 0 | 0
  Week 1 Moderate | 2 | 0 | 0 | 1
  Week 1 Severe | 0 | 0 | 0 | 0
  Week 1 Very Severe | 0 | 0 | 0 | 0
  Week 2 None | 26 | 34 | 15 | 16
  Week 2 Mild | 1 | 2 | 0 | 0
  Week 2 Moderate | 1 | 0 | 1 | 1
  Week 2 Severe | 0 | 0 | 0 | 0
  Week 2 Very Severe | 0 | 0 | 0 | 0
  Week 4 None | 22 | 32 | 13 | 16
  Week 4 Mild | 4 | 2 | 1 | 0
  Week 4 Moderate | 1 | 0 | 0 | 0
  Week 4 Severe | 0 | 0 | 0 | 0
  Week 4 Very Severe | 0 | 0 | 0 | 0
  Week 6 None | 24 | 33 | 11 | 14
  Week 6 Mild | 3 | 0 | 0 | 1
  Week 6 Moderate | 0 | 0 | 2 | 0
  Week 6 Severe | 0 | 0 | 0 | 0
  Week 6 Very Severe | 0 | 0 | 0 | 0
  ET None | 3 | 2 | 3 | 1
  ET Mild | 1 | 0 | 0 | 0
  ET Moderate | 1 | 0 | 0 | 1
  ET Severe | 2 | 0 | 0 | 0
  ET Very Severe | 0 | 0 | 0 | 0
  FUP None | 25 | 29 | 12 | 15
  FUP Mild | 1 | 1 | 1 | 0
  FUP Moderate | 1 | 0 | 1 | 1
  FUP Severe | 0 | 0 | 0 | 0
  FUP Very Severe | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Week 6
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | AD Vehicle Once Daily (QD) | AD PF-07038124 0.01% QD | Psoriasis Vehicle QD | Psoriasis PF-07038124 0.01% QD
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 6/34 | 1/36 | 6/17 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AD Vehicle Once Daily (QD) (N=34) | AD PF-07038124 0.01% QD (N=36) | Psoriasis Vehicle QD (N=17) | Psoriasis PF-07038124 0.01% QD (N=17)
Application site pruritus (General disorders) | 2 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT04664153/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04664153/SAP_001.pdf